CLINICAL TRIAL: NCT06269757
Title: Efficacy of an Individualized Exercise Program for Iliotibial Band Syndrome: A Randomized Controlled Study
Brief Title: Exercise Program for ITB Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01514
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Exercise Program (Experimental): Patients with diagnosed ITB syndrome indicated for non-operative management who are assigned to an individualized exercise program.
  Duration of therapy will be approximately 3 months. Patients will be followed for 6 months to assess longitudinal outcomes.
  Interventions: Behavioral: Individualized Exercise Program
- Standard Physical Therapy (Active Comparator): Patients with diagnosed ITB syndrome indicated for non-operative management who are assigned to receive standard physical therapy.
  Duration of therapy will be approximately 3 months. Patients will be followed for 6 months to assess longitudinal outcomes.
  Interventions: Behavioral: Standard Physical Therapy

INTERVENTIONS:
Behavioral: Individualized Exercise Program — The individualized exercise program involves an initial 2D individual running evaluation designed for runners of all ages and abilities, to help improve performance and prevent injury. During the assessment patients receive a one-on-one evaluation with an exercise physiologist that includes:
  * Running analysis;
  * Training program review;
  * Strength and flexibility assessment;
  * Review of running video;
  * Personalized final report.
  Arms: Individualized Exercise Program
Behavioral: Standard Physical Therapy — Standard of care physical therapy for ITB band syndrome involves exercises designed to target structural weaknesses such as hip abductor weakness. Typical exercises include but are not limited to hip flexor stretches, side lying hip abduction, figure 4 bridges, lateral walks with exercise bands, and side planks.
  Arms: Standard Physical Therapy

SUMMARY:
Patients with diagnosed iliotibial band (ITB) syndrome indicated for non-operative management will be randomized to individualized exercise program or standard physical therapy over the course of 3 months to determine any possible difference in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ITB syndrome
* Age 18-65
* Ability to comply with a standardized physical therapy protocol
* Willing and able to provide consent

Exclusion Criteria:

* Patients at any increased risk of falls or at increased risk from harm due to falling, including issues with vertigo, osteoporosis, or a history of past falls
* Patient otherwise deemed at increased risk from this investigational rehabilitation program by their referring surgeon or physical therapist
* Patients who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score Physical Short-Form (KOOS-PS) Score | Month 6
  The KOOS-PS4 contains seven items: rising from bed, putting on socks/stockings, rising from sitting, bending to floor, twisting/pivoting on your injured knee, kneeling and squatting. Participants indicate the degree of difficulty they face in performing the items, from "none" to "extreme." A final global score, from 0 (no problems) to 100 (extreme problems), is produced for the scale. Lower scores indicate greater physical function.
Visual Analogue Scale (VAS) Score | Month 6
  Pain is rated on a 10-point scale, from 0 (no pain) to 10 (worst possible pain). The total score is the response; lower scores indicate less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, MD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside of NYULH.